CLINICAL TRIAL: NCT02033317
Title: An Open-Label, Multiple Dose Study to Evaluate the Pharmacology, Safety, and Tolerability of Patiromer in Hemodialysis Patients
Brief Title: An Open-Label, Multiple Dose Study to Evaluate the Pharmacology, Safety, and Tolerability of Patiromer in Participants on Hemodialysis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to slow enrollment
Sponsor: Relypsa, Inc. (Industry)
Responsible Party: Sponsor
Organization: Vifor Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RLY5016-201
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — patiromer; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patiromer (Experimental)
  Interventions: Drug: patiromer

INTERVENTIONS:
Drug: patiromer — 15 grams/day (5 grams 3 times daily) administered orally
  Other Names: RLY5016 for Oral Suspension; Veltassa

SUMMARY:
This study assessed the pharmacodynamic effects of patiromer on serum potassium in participants on hemodialysis.

DETAILED DESCRIPTION:
The initial intent was to enroll 12-24 adult male and female participants on hemodialysis into the study. Due to significant recruitment challenges, the study was discontinued after six participants were enrolled in the study.

This was an open-label, multiple-dose, adaptive-design study in participants on hemodialysis. Eligible participants on hemodialysis were to remain in the Clinical Research Unit for 2 weeks (Day -7 to Day 8) and were required to consume a potassium, magnesium, calcium and sodium-controlled diet.

ELIGIBILITY:
Inclusion Criteria:

* Participants on hemodialysis between the ages of 18 and 70 years, with serum potassium levels of at least 5.5 mmol/L
* Adequately dialyzed (Kt/V ≥ 1.2)

Exclusion Criteria:

* History of bowel obstruction, swallowing disorders, severe gastrointestinal disorders or major gastrointestinal surgery.
* Severe constipation or irregular bowel habits.
* Unable to consume or tolerate the study-specific diet.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Development, Study Director — Relypsa, Inc.
Locations (2):
- United States (2):
  - Investigator Site, Orlando, Florida
  - Investigator Site, Minneapolis, Minnesota

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study population consisted of participants on hemodialysis between the ages of 18 and 70 years, with pre-dialysis serum potassium levels of at least 5.5 mmol/L prior to the study.
Groups:
- Patiromer: 15 grams/day (5 grams 3 times daily) patiromer administered orally
Period: Overall Study
Arm/Group | Patiromer
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patiromer
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 49.7 [44 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Potassium (Day 1 to Day 8)
Time Frame: Day 1 and Day 8
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Patiromer
Number analyzed (Participants) | 6
mmol/L | -0.23 (0.327)
Statistical Analysis 1: Comparison: Patiromer; Test type: Superiority or Other; p = 0.14, paired t-test

2. Primary Outcome: Change From Baseline in Fecal Potassium Excretion (Day -7 Through Day -1) and Treatment (Day 1 Through 7)
Time Frame: Day -7 Through Day -1 and Day 1 Through Day 7
Measure: Mean (Standard Deviation); unit: mg/Day
Arm/Group | Patiromer
Number analyzed (Participants) | 6
mg/Day | 359 (277)
Statistical Analysis 1: Comparison: Patiromer; Test type: Superiority or Other; p = 0.02, paired t-test

ADVERSE EVENTS:
Time Frame: Up to 10 days after Day 8 or last patiromer dose, whichever was earlier.
Description: Participants who received at least one dose of trial medication.
Arm/Group | Patiromer
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patiromer (N=6)
Abdominal Rigidity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Furuncle (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
The initial intent was to enroll 12-24 adult male and female participants on hemodialysis into the study. Due to significant recruitment challenges, the study was discontinued after six participants were enrolled in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreements generally provide that PI cannot publish single site data before publication of the multi-site publication, unless 1 year has elapsed since completion of the study at all sites. Thereafter, PI may publish provided that PI shall: provide a copy of the publication to sponsor at least 60 days in advance of submission for publication; delete sponsor's confidential information as requested; and delay publication up to an additional 90 days to permit protection of intellectual property.